CLINICAL TRIAL: NCT06916949
Title: The Role of High-fidelity Medical Simulation in Managing Emotional Components and Stress During Emergency and Urgent Care
Brief Title: Stress Evaluation and Management Using High Fidelity Simulation in Medical Education
Acronym: STRATAGEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID7328
Record Dates: First submitted 2025-02-11; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-01

CONDITIONS: Stress; Pupillometry; High Fidelity Simulation Training; Resident Education; Heart Rate Variability, Biomarker of Stress; Simulation Training
MeSH Terms: interventions — Electrocardiography; Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulation team (Experimental): All participants will be divided in teams, each one consisting of three medical trainees from the same specialty training program, and all of them will undergo two high-fidelity simulations based on a clinical scenario relevant to their specialization.
  Interventions: Diagnostic Test: Electrocardiogram; Diagnostic Test: Pupillometry; Diagnostic Test: Electroencephalogram

INTERVENTIONS:
Diagnostic Test: Electrocardiogram — two leads ECG
  Other Names: ECG, EKG
Diagnostic Test: Pupillometry — During the simulation, automatic pupillometry will be performed on all team members at the following time points: Baseline (T0) During the simulation (T1) End of the simulation (T2) End of the debriefing (T3)
Diagnostic Test: Electroencephalogram — EEG monitoring throughout the entire simulation. The EEG recordings will be sampled at: Baseline (T0) During the simulation (T1) End of the debriefing (T2)
  Other Names: EEG

SUMMARY:
The goal of this interventional study is to collect clinical and neurophysiological information to determine whether high-fidelity simulation can serve as a stress-inducing stimulus in a population of healthy residents (Emergency medicine, Anesthesia and Intensive care medicine, Paediatrics), both male and female, aged between 25 and 40 years. The main questions it aims to answer are:

1. Define in which phase of the simulation the highest level of stress is observed.
2. Determine the level of stress reached after performing a second high-fidelity simulation after a period of time.
3. Identify whether specific brain areas are activated during high-fidelity simulation.

Participants will form teams, consisting of three medical trainees from the same specialty training program, that will undergo two high-fidelity simulations based on a clinical scenario relevant to their residency.

* During the simulation, automatic pupillometry will be performed on all team members at the four time points.
* Additionally, a two-lead ECG will be recorded for all team members at baseline and end of the debriefing
* One team member will undergo EEG monitoring throughout the entire simulation. The EEG recordings will be sampled at baseline, during the simulation and end of the debriefing.

ELIGIBILITY:
Inclusion Criteria:

* Medical trainees from the specialties of Emergency Medicine, Anesthesia and Intensive Care, Clinical Toxicology, Pediatrics, and Neonatology.
* Normal hearing and vision, or corrected to normal.

Exclusion Criteria:

* Known history of psychiatric disorders, cognitive impairment, or cardiac arrhythmias.
* Current treatment with psychoactive, cardio-stimulant, or cardio-inhibitory medications.
* Significant stressful life events in the past six months (e.g., family bereavement).
* Previous systematic experience in meditation.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) Analysis in the time domain | From the enrolment to two weeks after
  To assess whether stress levels vary during simulation phases. All subjects will undergo electrocardiographic (ECG) recording at baseline and at the end of the debriefing using a portable Holter ECG device. The ECG traces will then be extracted, artifact-cleaned, and converted for Heart Rate Variability (HRV) analysis using dedicated software. HRV is a measure of the variation in R-R intervals between consecutive heartbeats and reflects the extrinsic regulation of heart rate mediated by the autonomic nervous system on the sinoatrial node.
Heart rate variability (HRV) analysis in the frequency domain | from the enrolment to two weeks after
  Low frequency (LF) reflects the simultaneous influence of both sympathetic and parasympathetic control on the sinoatrial node; and high frequency (HF) reflects parasympathetic nervous system modulation.
  The LF/HF ratio will be calculated as an indicator of the sympathovagal balance.

SECONDARY OUTCOMES:
Changes in autonomic parameters in response to stress induced by high-fidelity simulation: automatic pupillometry. | From the enrolment to two weeks after
  The subjects undergo quantitative measurement of the pupillary light reflex at four time points: baseline, during simulation, at the end of the simulation, and at the end of the debriefing. The technique involves exposing both pupils of the subjects to an infrared light stimulus and assessing their reactivity parameters using an infrared sensor. The instrument used for data collection is the NPi-200 (NeurOptics, Irvine, CA, USA), a portable pupillometer that provides a light stimulus with fixed intensity (1000 lux) and duration (0.8s). We measure the Neurological Pupillary Index (NPI), a composite parameter, automatically derived, indicative of pupillary reactivity. An NPi ≥ 3 is considered normal.
Identify brain areas involved during simulation using EEG | From the enrolment to two weeks after
  Identify whether specific brain areas are activated during high-fidelity simulation.
  One member from each simulation team (identified as the team leader) will undergo continuous electroencephalographic (EEG) monitoring using a 19-electrode device in fixed positions according to the international 10-20 system during three phases of the advanced medical simulation:
  * Baseline stage during quiet wakefulness (eyes closed);
  * During the medical simulation;
  * During the debriefing. The EEG recordings will be transmitted to a computer and analyzed using the eLORETA software (exact Low Resolution Brain Electromagnetic Tomography), that allows connectivity analysis. The study of brain connectivity allows for the identification of statistically significant synchronization between signals recorded from two or more electrodes. Connectivity can be estimated as functional connectivity, which is bidirectional and does not determine a causal effect.
Variation of stress level over time using Perceived Stress Scale 10 | From the enrolment to two weeks after
  Determine the level of stress reached after performing a second high-fidelity simulation after a period of time.
  Assessment of Stress Level and Emotional Component through the completion of the Perceived Stress Scale 10 (PSS-10) by the medical trainee. This scale consists of ten items, with each item rated on a scale from 0 (not stressful at all) to 4 (very stressful), focusing on thoughts and emotions experienced over the past 30 days.
  A score between 0 and 13 indicates good emotional management in both personal and professional life.
  A score between 14 and 26 suggests initial difficulties in managing emotions and stress.
  A score between 27 and 40 indicates an excessive stress load that negatively affects the individual's well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gullì, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: All researchers that wish to, can gain access to the IPD and supporting information by contacting the corresponding author

REFERENCES:
- [Background] Champeroux P, Fesler P, Jude S, Richard S, Le Guennec JY, Thireau J. High-frequency autonomic modulation: a new model for analysis of autonomic cardiac control. Br J Pharmacol. 2018 Aug;175(15):3131-3143. doi: 10.1111/bph.14354. Epub 2018 Jun 15. PMID 29723392
- [Background] Niskanen JP, Tarvainen MP, Ranta-Aho PO, Karjalainen PA. Software for advanced HRV analysis. Comput Methods Programs Biomed. 2004 Oct;76(1):73-81. doi: 10.1016/j.cmpb.2004.03.004. PMID 15313543